CLINICAL TRIAL: NCT02749006
Title: A Randomized Double-blind Sham-controlled Trial of Repetitive Transcranial Magnetic Stimulation (rTMS) in Acute Bipolar Depression
Brief Title: Efficacy of rTMS in Bipolar Depression
Acronym: rTMS-BD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll the planned number of participants.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lakshmi N Yatham, Prinicipal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H16-00259
Record Dates: First submitted 2016-03-18; First posted 2016-04-22 (Estimated); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Bipolar Depression
Keywords: Bipolar disorder; Depression; intermittent Theta-Burst Stimulation (rTMS); neuromodulatory technique
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active iTBS rTMS (Active Comparator): The active arm involves magnetic stimulation of the brain to the left dorsolateral prefrontal cortex (DLPFC) daily for four weeks. The active arm will be receiving intermittent Theta-Burst (iTBS) repetitive Transcranial Magnetic Stimulation (rTMS) to deliver magnetic pulses.
  Interventions: Device: iTBS repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham rTMS (Sham Comparator): sham rTMS treatment involves scalp stimulation with no magnetic pulse daily for four weeks (20 sessions). Sham rTMS involves only the click replicating the sound of the magnetic discharge, without any magnetic pulse being delivered.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: iTBS repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS is a non-invasive procedure in which cerebral electrical activity is influenced by a rapidly changing magnetic field. The magnetic field is created by a plastic-encased coil which is placed over the patient's scalp. The magnetic field can be directed onto specific areas of the brain. rTMS can modulate cerebral activity by low or high frequencies. Over time, the magnetic field pulses can gradually change the activity level of the stimulated brain region and help symptoms of bipolar depression.
  Other Names: MAGPRO X100 stimulator
  Arms: Active iTBS rTMS
Device: Sham rTMS — Sham rTMS involves a click replicating the sound of the magnetic discharge, without any magnetic pulse being delivered.
  Other Names: MAGPRO X100 stimulator
  Arms: Sham rTMS

SUMMARY:
Bipolar Disorder is a common condition that is characterized by periods of mood elevation however periods of chronic and recurring depressive episodes are more common and can be severely disabling. Effective treatments exist, however a significant portion of bipolar depressed patients do not respond to, or have difficulty tolerating many of these interventions. Repetitive Transcranial Magnetic Stimulation (rTMS) is a non-invasive neuromodulatory technique that is effective in major depression and there is evidence for its efficacy in bipolar depression which needs to be assessed in larger randomized controlled trials. This study is a randomised, double-blind, sham-controlled trial over four weeks. The primary objective is to assess improvement in depressive symptoms in acute bipolar depressed patients on treatment with intermittent Theta-Burst Stimulation (iTBS) in comparison to sham-rTMS.

DETAILED DESCRIPTION:
rTMS is a treatment that involves stimulating a certain area of the brain with magnetic field pulses. Over time, the magnetic field pulses can gradually change the activity level of the stimulated brain region and help symptoms of bipolar depression. The device used in this study has been approved by Health Canada for therapeutic use since 2002. Participants will complete a screen visit to determine eligibility based on the inclusion/exclusion criteria. If the participants are not eligible, no further study procedures will be conducted. Eligible subjects will be randomized to receive either active iTBS-rTMS or sham rTMS treatment (scalp stimulation with no magnetic pulse) daily for four weeks (20 sessions) to the left dorsolateral prefrontal cortex (DLPFC). All participants will complete a MRI (to target the left DLPFC region of the brain and functional activity), EEG & fNIRS, lab work, and neurocognitive testing prior to the commencement and post rTMS treatment. Efficacy, safety and tolerability will be evaluated at screen visit, during daily rTMS treatments, clinic visits and post rTMS treatment. All participants will have a phone interview two weeks post rTMS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Are a male or female aged 18 to 70 years.
* Have a diagnosis of Bipolar Disorder with a current ongoing episode of depression.
* Are not currently experiencing a mania.
* Have failed to achieve a clinical response or have been unable to tolerate an adequate dose of at least one of the medications used for treating Bipolar depression
* Are taking an anti-manic agent (lithium or valproate) or an atypical antipsychotic (quetiapine, lurasidone, aripiprazole, ziprasidone, risperidone, olanzapine), or a combination of the above, or a combination of any of them with lamotrigine 100-400 mg daily. Lamotrigine alone for bipolar II disorder is permitted.
* current medications have been at a stable dose in the 2 weeks prior to randomization
* Are capable of understanding, consenting to, and complying with the requirements of the study

Exclusion criteria:

* Have an alcohol or substance abuse or dependence within the last 3 months.
* Are at a significant risk of harm to themselves or others
* Are pregnant or planning on becoming pregnant in near future or lactating.
* Have a personal or family history of seizures.
* Have a history of unstable or inadequately treated medical illnesses, including moderate to severe brain injury or head trauma.
* Have a primary diagnosis of other psychiatric disorders (other than Bipolar) or personality disorders that are of primary concern and causing greater impairment other than bipolar disorder.
* are currently taking more than 3 of the antipsychotics.
* Have failed a course of ECT in the current episode.
* History of non-response to rTMS treatment.
* If participating in psychotherapy, you must have been in stable treatment for at least 3 months prior to entry into the study,
* Currently (or in the last 4 weeks) taking more than 2 mg daily (or equivalent) of lorazepam or any dose of medication for seizures
* Have a pacemaker, or an implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth that cannot be safely removed.
* Have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Yatham, MBBS,FRCPsy, Study Director — Regional Head and Program Medical Director,
Locations (2):
- Canada (2):
  - Dr. Alexander McGirr, Calgary, Alberta
  - Djavad Mowfaghian Centre for Brain Heath, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torres IJ, Ge R, McGirr A, Vila-Rodriguez F, Ahn S, Basivireddy J, Walji N, Frangou S, Lam RW, Yatham LN. Effects of intermittent theta-burst transcranial magnetic stimulation on cognition and hippocampal volumes in bipolar depression. Dialogues Clin Neurosci. 2023 Dec;25(1):24-32. doi: 10.1080/19585969.2023.2186189. PMID 36924413
- [Derived] McGirr A, Vila-Rodriguez F, Cole J, Torres IJ, Arumugham SS, Keramatian K, Saraf G, Lam RW, Chakrabarty T, Yatham LN. Efficacy of Active vs Sham Intermittent Theta Burst Transcranial Magnetic Stimulation for Patients With Bipolar Depression: A Randomized Clinical Trial. JAMA Netw Open. 2021 Mar 1;4(3):e210963. doi: 10.1001/jamanetworkopen.2021.0963. PMID 33710288

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by referral, as well as online and community advertisements 2 Canadian centers (University of British Columbia [UBC], British Columbia, Canada; and University of Calgary [UC], Alberta, Canada) between October 2016 and March 2020 .
Pre-assignment Details: Of the 71 assessed for eligibility 37 were randomized.
Period: Overall Study
Arm/Group | Active iTBS rTMS | Sham rTMS
Started | 18 | 19
Completed | 15 | 16
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active iTBS rTMS | Sham rTMS | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.78 (13.71) | 43.00 (14.34) | 43.86 (13.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 18 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Primary Diagnosis [Count of Participants; unit: Participants]
  Bipolar disorder type I | 11 | 10 | 21
  Bipolar disorder type II | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS) Scale Score
Description: The primary outcome was the change in score on the Montgomery-Asberg Depression Rating Scale from baseline to study end. A higher score means a worse outcome. Min value is 0, Max value is 60
Time Frame: Baseline, Week 2, Week 4
Population: Diagnosis of BD type I or type II by Diagnostic and Statistical Manual of Mental Disorders (Fifth Edition) criteria, experiencing a major depressive episode (MDE).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active iTBS rTMS | Sham rTMS
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 32.27 (4.04) | 31.52 (5.22)
  Week 2: number analyzed (Participants) | 16 | 17
  Week 2 | 24.12 (10.09) | 25.17 (8.24)
  Week 4: number analyzed (Participants) | 15 | 16
  Week 4 | 24.46 (10.82) | 23.06 (10.58)

2. Secondary Outcome: Number of Participants With Clinical Response
Description: Response rates are defined as patients showing ≥50% reduction in MADRS scores.
Time Frame: Baseline to Week 4 (assessed at Week 2 and Week 4, Week 4 reported)
Measure: Count of Participants; unit: Participants
Arm/Group | Active iTBS rTMS | Sham rTMS
Number analyzed (Participants) | 18 | 19
Participants | 3 | 3

3. Secondary Outcome: Number of Participants Meeting Criteria for Clinical Remission
Description: Clinical Remission is defined as a MADRS score ≤12
Time Frame: Baseline to Week 4 (assessed at Week 2 and Week 4, Week 4 reported)
Measure: Count of Participants; unit: Participants
Arm/Group | Active iTBS rTMS | Sham rTMS
Number analyzed (Participants) | 18 | 19
Participants | 3 | 3

4. Secondary Outcome: Overall Well Being
Description: The visual analog scale (VAS) is a self report measure that captures the over all well being. Min 0-worse health to Max 100- best health.
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active iTBS rTMS | Sham rTMS
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 41.83 (18.29) | 35.21 (18.80)
  Week 4 | 58.13 (17.13) | 46.66 (18.09)

5. Secondary Outcome: Brief Illness Perception Questionnaire
Description: Brief Illness Perception Questionnaire measures participant's perception of illness. Min = 0 Max = 80. Higher score means worse outcome.
Time Frame: Baseline to 4 weeks
Population: Not all participants completed the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active iTBS rTMS | Sham rTMS
Number analyzed (Participants) | 17 | 18
score on a scale
  Baseline | 60.35 (4.67) | 59.13 (8.21)
  Week 4: number analyzed (Participants) | 16 | 15
  Week 4 | 57.31 (8.27) | 58.93 (8.37)

6. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: The Sheehan Disability Scale is a five-item, self-rated questionnaire designed to measure the extent to which a patient's disability due to an illness interferes with work/school, social life/leisure activities, and family life/home responsibilities. Each subscale score (a work disability, a social life disability, a family life disability) is combined into a single total score (sum of the non missing responses for items 1-3) representing a global impairment rating, ranging from 0 to 30, with higher scores indicative of significant functional impairment.
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active iTBS rTMS | Sham rTMS
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 23.83 (5.09) | 23.44 (6.43)
  Week 4 | 19.40 (10.32) | 19.23 (8.26)

7. Secondary Outcome: Quality of Life Questionnaire
Description: The Quality of Life in Bipolar Disorder scale is a 56 item scale which assesses 12 core and 2 optional (work and study) domains, each containing four self-report items (1: strongly disagree to 5: strongly agree). An overall score (range: 48-240) may be calculated by summing responses to the 48 items of the core 12 domains. Higher scores reflect greater satisfaction with a person's quality of life.
Time Frame: Baseline to 4 weeks
Population: Not all participants completed the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active iTBS rTMS | Sham rTMS
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 109 (18.67) | 108.78 (26.34)
  Week 4: number analyzed (Participants) | 16 | 13
  Week 4 | 136.18 (33.81) | 130.76 (36.54)

8. Secondary Outcome: Patient Global Impression Rating Scale: Severity
Description: Patient Global Impression Rating Scale: Severity rates how depressed the participant is at the current time. 1-4 (1 is normal and 4 is severe)
Time Frame: Baseline to 4 weeks
Population: Not all participants completed the scale at Week 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active iTBS rTMS | Sham rTMS
Number analyzed (Participants) | 18 | 18
score on a scale
  Baseline | 3.16 (0.51) | 3.05 (0.80)
  Week 4: number analyzed (Participants) | 15 | 15
  Week 4 | 2.60 (0.82) | 2.66 (0.81)

9. Secondary Outcome: Patient Global Impression Rating Scale- Improvement
Description: Rates current depression compared to baseline. Min =1 Max =7 Higher scores mean worse outcome.
Time Frame: Week 4
Population: Not all participants completed the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active iTBS rTMS | Sham rTMS
Number analyzed (Participants) | 15 | 15
score on a scale | 3.53 (1.24) | 3.20 (1.26)

ADVERSE EVENTS:
Time Frame: Baseline to 4 weeks
Description: Systematic collection of Non-Serious Adverse events occurred only at the DMCBH site in Vancouver.
Arm/Group | Active iTBS rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 7/7 | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active iTBS rTMS (N=7) | Sham rTMS (N=9)
Pain and discomfort at treatment site (Nervous system disorders) | 4 (4) | 2 (2)
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 4 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 5 (5) | 4 (4)
Stomach Cramp/ Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
This study is limited by a modest sample size; however, this is the direct consequence of premature termination after interim analyses indicated futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT02749006/Prot_SAP_000.pdf